CLINICAL TRIAL: NCT02310100
Title: TactiCath® Contact Force Ablation Catheter Study for Atrial Fibrillation Post Approval Study
Acronym: TactiCathPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10030; NCT02088606 (obsolete NCT alias)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TactiCath Quartz (Experimental): TactiCath Quartz treatment
  Interventions: Device: TactiCath Quartz treatment

INTERVENTIONS:
Device: TactiCath Quartz treatment

SUMMARY:
A prospective, multicenter, interventional study to collect confirmatory evidence on the safety and effectiveness of the TactiCath® percutaneous ablation catheter in the post approval setting for the treatment of symptomatic paroxysmal atrial fibrillation using contact force assisted irrigated radiofrequency ablation.

DETAILED DESCRIPTION:
The TactiCath Quartz PAS is a prospective, non-randomized, multicenter, interventional study to evaluate the continued safety and effectiveness of the TactiCath Quartz Set for the treatment of symptomatic paroxysmal atrial fibrillation (PAF) using contact force assisted irrigated RF ablation.

Patients undergoing elective catheter ablation for symptomatic PAF who are refractory or intolerant to at least one antiarrhythmic drug (Class I-IV) will be screened for enrollment. Patients who meet the study entry criteria and sign the patient informed consent form will be enrolled and treated following the standard of care at each study site.

After the index procedure, subjects will be followed for a total of 60 months. During the 3-month blanking period following ablation, subjects may undergo up to 2 repeat ablation procedures (up to 10 days prior to end of the blanking period) using the same device used during ablation. Subjects will be evaluated at pre-discharge, at 7 days, at 3, 6 and 12 months post-index procedure and then yearly thereafter. Subjects will complete Holter monitoring at 3- and 6- months post index ablation procedure and at yearly intervals beginning at 12 months post-index ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is planned to undergo a catheter ablation procedure due to symptomatic PAF that is refractory or intolerant to at least one Class I IV antiarrhythmic drug
2. Minimum of one episode of PAF greater than 30 seconds in duration within 12 months prior to enrollment documented by 12 lead electrocardiogram (ECG), Holter monitor, trans-telephonic event monitor, telemetry strip, or implanted device
3. Minimum of 3 episodes of PAF within the preceding 12 months documented by patient history
4. Patient is 18 years of age or older
5. Patient is willing and capable of complying unassisted with the study protocol requirements including all specified follow up visits
6. Patient provides written informed consent prior to enrollment in the study

Exclusion Criteria:

1. Persistent or long-standing persistent atrial fibrillation (AF)
2. Patient has had 4 or more cardioversions in the past 12 months.
3. Active systemic infection
4. Presence of implantable cardiac defibrillator (ICD)
5. Arrhythmia due to reversible causes including thyroid disorders, acute alcohol intoxication, and other major surgical procedures in the preceding 3 months
6. Myocardial infarction (MI), acute coronary syndrome, percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery within preceding 3 months
7. Left atrial diameter > 5.0 cm
8. Left ventricular ejection fraction < 35%
9. New York Heart Association (NYHA) class III or IV
10. Previous left atrial ablation procedure, either surgical or catheter ablation
11. Patient has had a left atrial surgical procedure or incision with resulting scar
12. Previous tricuspid or mitral valve replacement or repair
13. Heart disease in which corrective surgery is anticipated within 6 months
14. Bleeding diathesis or suspected pro coagulant state
15. Contraindication to long term antithromboembolic therapy
16. Presence of any condition that precludes appropriate vascular access
17. Renal failure requiring dialysis
18. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
19. Contraindication to computed tomography and magnetic resonance angiography
20. Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
21. Positive pregnancy test results for female patients of childbearing potential
22. Patient has other anatomic or co morbid conditions that, in the investigator's opinion, could limit the patient's ability to participate in the study or to comply with follow up requirements, or impact the scientific soundness of the study results
23. Patient is currently participating in another clinical trial or has participated in a clinical trial within 30 days prior to screening that may interfere with this study
24. Patient is unlikely to survive the protocol follow up period of 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, PhD, Study Director — Abbott
Locations (20):
- United States (20):
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Regional Cardiology Associates, Sacramento, California
  - Emory University Hospital, Atlanta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Cardiology Consultants of East Michigan, Flint, Michigan
  - Providence Hospital, Southfield, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Mount Sinai Hospital, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 109 subjects were directly enrolled into the TactiCath PAS 50 subjects rolled over from the TactiCath Continued Access Protocol 19 subjects rolled over from the TOCCASTAR Supplemental Study The first subject was enrolled on January 21, 2015 and the last subject on January 29, 2016.
  All enrollment was from sites within the United States.
Pre-assignment Details: Only subjects that met all inclusion criteria and did not meet any exclusion criteria were enrolled in the study.
Groups:
- TactiCath Quartz: Patients undergoing elective catheter ablation for symptomatic paroxysmal AF that was refractory or intolerant to at least one Class I-IV antiarrhythmic drug
Period: Overall Study
Arm/Group | TactiCath Quartz
Started (FDA approval) | 178 (First enrollment)
Completed | 160
Not Completed | 18
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 10
Not completed — Enrollment closure | 1
Not completed — Unapproved ablation operator | 1
Not completed — Visit compliance | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Patient demographics and baseline characteristic variables were summarized descriptively by treatment group.
Groups:
- TactiCath Quartz: Ablation with TactiCath Quartz
Arm/Group | TactiCath Quartz
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 subjects had missing data for sex
  Participants
    Sex: number analyzed (Participants) | 176
    Sex: Female | 73
    Sex: Male | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 176
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 172
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 178

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Recurrent, Symptomatic Paroxysmal Atrial Fibrillation (PAF), Atrial Flutter (AFL), and Atrial Tachycardia (AT)
Description: Rate of subjects free from symptomatic Paroxysmal Atrial Fibrillation (PAF), Atrial Flutter (AFL), and Atrial Tachycardia (AT) lasting longer than 30 seconds through 9 months of follow-up after a 3 month blanking period compared to a stated performance goal. Procedural failure defined by any of the following events: (1) Documented recurrence of AF/AFL/AT during the 9-month observational period lasting longer than 30 seconds; (2) Repeat ablation following the blanking period; or (3) Use of s new anti-arrhythmic drug for the documented symptomatic atrial arrhythmia following the blanking period.
Time Frame: 12 Months post ablation
Population: Subjects who terminated the study prematurely before experiencing a treatment failure were not considered a treatment success at 12-months. Subjects who terminated the study for reasons clearly unrelated to the study device were also excluded and not considered treatment failures.
Measure: Count of Participants; unit: Participants
Groups:
- TactiCath Quartz: Ablation using TactiCath Quartz
Arm/Group | TactiCath Quartz
Number analyzed (Participants) | 165
Participants | 111
Statistical Analysis 1: Comparison: TactiCath Quartz; H0: PE ≤ 54.9% Ha: PE > 54.9% Where PE is the primary effectiveness endpoint rate; Test type: Other — This is a one-group comparison to a performance goal; p = 0.0008, Exact binomial; binomial proportion = 0.673, 95% CI 1-sided [lower limit 0.608]

2. Primary Outcome: Number of Participants Experiencing a Device or Procedure-related Serious Adverse Event
Description: The rate of device or procedure serious adverse events occurring within 7 days of the index procedure or hospital discharge, whichever is later, compared to a stated performance goal.
Time Frame: 7 days
Population: The analysis population includes all subjects in whom a study device was introduced.
Measure: Count of Participants; unit: Participants
Arm/Group | TactiCath Quartz
Number analyzed (Participants) | 173
Participants | 14
Statistical Analysis 1: Comparison: TactiCath Quartz; H0: PS ≥ 16.2% Ha: PS < 16.2% where PS is the primary safety endpoint rate; Test type: Other — One group comparison to a performance goal; p = 0.0013, Exact binomial; binomial proportion = 0.081, 95% CI 1-sided [upper limit 0.124]

ADVERSE EVENTS:
Time Frame: 2 years
Description: -NOTE: 5 subjects withdrew before the TactiCath Quartz catheter was introduced into the body resulting in a denominator of 173 in this section.
  Investigators reported all AEs except for the following:
  * Exacerbation of pre-existing non-CV conditions
  * Physical trauma unrelated to the procedure
  * New disease unrelated to AF, the procedure, or study device/CV drugs
  * Common ailments unrelated to the CV system, the procedure, study device or drugs used to treat CV illness
Arm/Group | TactiCath Quartz
All-Cause Mortality (participants affected / at risk) | 0/173
Serious Adverse Events (participants affected / at risk) | 14/173
Other Adverse Events (participants affected / at risk) | 30/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TactiCath Quartz (N=173)
Vascular access complication (Surgical and medical procedures) | 5 (5)
Cardiac perforation/tamponade (Cardiac disorders) | 4 (4)
Hospitalization (General disorders) | 4 (4)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Allergic drug reaction that required intubation (General disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TactiCath Quartz (N=173)
Chest pain (General disorders) | 8 (8)
Other (General disorders) | 14 (14)
Pericarditis (Cardiac disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02310100/Prot_SAP_000.pdf